CLINICAL TRIAL: NCT01953731
Title: A Phase 1, Open-Label Fixed-Sequence 2-Period Study To Investigate The Effect Of Multiple Doses Of Rifampin On Palbociclib (PD-0332991) Pharmacokinetics In Healthy Volunteers
Brief Title: A Study To Investigate The Drug-Drug Interaction Potential Of Rifampin OnThe Investigational Agent Palbociclib (PD-0332991)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A5481017
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
Keywords: palbociclib; PD-0332991; rifampin; drug-drug interaction study
MeSH Terms: interventions — palbociclib; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-Arm Fixed-Sequence (Experimental): Subjects will receive two different interventions in fixed-sequence two-period study. In the first period the subjects will receive a single-dose of palbociclib. In the second period, subjects will receive 12 days of rifampin and a single dose of palbociclib on day 8. In both periods, subjects will undergo pharmacokinetic sampling at prespecified time points up to 120 hours post palbociclib dose.
  Interventions: Drug: Palbociclib; Drug: Rifampin

INTERVENTIONS:
Drug: Palbociclib — In period 1, patients will receive a single 125mg oral dose of palbociclib alone. Subjects will undergo palbociclib pharmacokinetic sampling at prespecified time points up to 120 hours post palbociclib dose.
  In period 2, subjects will receive 12 daily oral doses of 600mg of rifampin and a single 125mg oral dose of palbociclib on day 8. Subjects will undergo palbociclib pharmacokinetic sampling at prespecified time points up to 120 hours post palbociclib dose.
  Other Names: palbociclib, PD-0332991
Drug: Rifampin — In period 2, subjects will receive 12 daily oral doses of 600mg of rifampin and a single 125mg oral dose of palbociclib on day 8. Subjects will undergo palbociclib pharmacokinetic sampling at prespecified time points up to 120 hours post palbociclib dose.
  Other Names: palbociclib, PD-0332991, rifampin, rifampicin

SUMMARY:
This study will compare the plasma pharmacokinetics of a single 125mg oral dose of palbociclib in the presence and absence of rifampin-mediated enzyme induction in a fixed-sequence two-period study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females of non-childbearing potential
* body mass index between 17.5-30.5 kg/m2 with a total body weight greater than 50kg

Exclusion Criteria:

* Evidence or history of any clinically significant physiologic, psychological, or medical conditions
* a positive drug screen or alcohol breath test
* a baseline ECG demonstrating a QTc>450msecs or a QRS interval >120msecs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 0-120 hours post-dose
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Maximum Observed Plasma Concentration (Cmax) | 0-120 hours post-dose

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0-120 hours post-dose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0-120 hours post-dose
Plasma Decay Half-Life (t1/2) | 0-120 hours post-dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent Oral Clearance (CL/F) | 0-120 hours post-dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) | 0-120 hours post-dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481017&StudyName=A%20Study%20To%20Investigate%20The%20Drug-Drug%20Interaction%20Potential%20Of%20Rifampin%20OnThe%20Investigational%20Agent%20Palbociclib%20%28PD-0332991%29%0A